CLINICAL TRIAL: NCT03118024
Title: Perioperative Management of Deep Inferior Epgastric Perforator (DIEP) Flap for Breast Reconstruction
Brief Title: Perioperative Management of DIEP Flaps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Dr. Alexandra Anker, Principal Investigator, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-101-0293
Record Dates: First submitted 2017-03-25; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Mammaplasty; Microsurgery; Free Tissue Flaps
Keywords: deep inferior epigastric perforator flap; fluid restriction; catecholamine restriction
MeSH Terms: interventions — Crystalloid Solutions; Catecholamines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid restriction (Active Comparator): Crystalloid fluid max. 2.0 ml/kg/h, no administration of colloids, noradrenaline max. 0.15 µg/kg/min
  Interventions: Drug: Crystalloid Solutions
- Catecholamine restriction (Active Comparator): Noradrenaline max. 0.04 µg/kg/min, fluids max. 8.0 ml/kg/h
  Interventions: Drug: Catecholamines

INTERVENTIONS:
Drug: Crystalloid Solutions — crystalloid restrictive anesthesia protocol
  Arms: Fluid restriction
Drug: Catecholamines — catecholamine restrictive anesthesia protocol
  Other Names: Norephinephrine
  Arms: Catecholamine restriction

SUMMARY:
By comparison of two different protocols with diverse fluid/ catecholamine administration limits (fluid restriction vs. catecholamine restriction with target systolic blood pressure > 100 mmHg) the investigators would like to reveal the impact of intraoperative blood pressure management on the survival rate of free deep inferior epigastric artery flaps for breast reconstruction.

ELIGIBILITY:
Inclusion criteria:

* Informed consent for study participation
* Every patient undergoing breast reconstruction (primary and secondary reconstruction) with deep inferior epigastric perforator flap at our hospital is offered to participate in the study

Exclusion criteria:

* No informed consent for study participation
* Patients with a high thromboembolic risk profile
* During pregnancy and breastfeeding
* Minors
* Patients with a health care proxy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Free flap survival rate | 5 days postoperatively
  Rates of (partial) flap loss in each study arm

SECONDARY OUTCOMES:
Period of hospitalization | up to 14 days
  Length of postoperative hospitalization in each study arm

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eley KA, Young JD, Watt-Smith SR. Epinephrine, norepinephrine, dobutamine, and dopexamine effects on free flap skin blood flow. Plast Reconstr Surg. 2012 Sep;130(3):564-570. doi: 10.1097/PRS.0b013e31825dbf73. PMID 22929242
- [Background] Motakef S, Mountziaris PM, Ismail IK, Agag RL, Patel A. Emerging paradigms in perioperative management for microsurgical free tissue transfer: review of the literature and evidence-based guidelines. Plast Reconstr Surg. 2015 Jan;135(1):290-299. doi: 10.1097/PRS.0000000000000839. PMID 25539313